CLINICAL TRIAL: NCT05208320
Title: Effectiveness of Community Health Workers in Hypertension Adherence: a Community Intervention in Elderly Patients
Brief Title: Effectiveness of Community Health Workers in Hypertension Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pham Ngoc Thach University of Medicine (Other)
Responsible Party: Principal Investigator, Cao Nguyen Hoai Thuong, Lecturer, Pham Ngoc Thach University of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8286
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention ward (Experimental): Patients received interventions as follow:
  * The health education syllabus included 4 chapters: (1) introduction to hypertension, (2) complications of high blood pressure, (3) lifestyle management, and (4) SCORE - European High-Risk Chart
  * Home health education by Community Health Workers every month for 6 months
  Interventions: Behavioral: Adherence
- control ward (No Intervention): Patients received usual care, consisted of existing services in the community

INTERVENTIONS:
Behavioral: Adherence — Patients received interventions as follow:
  * The health education syllabus included 4 chapters: (1) introduction to hypertension, (2) complications of high blood pressure, (3) lifestyle management, and (4) SCORE - European High-Risk Chart
  * Home health education by Community Health Workers every month for 6 months
  Arms: intervention ward

SUMMARY:
A community intervention in elderly hypertension patients by Community Health Workers in order to improve patients adherence to treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 60 years and older who had been diagnosed with hypertension for more than 3 months at the time of the study were eligible for inclusion.

Exclusion Criteria:

* People who are not able to answer interviews or have mental illnesses.
* Those who, after being interviewed, re-confirmed that they did not have a diagnosis of hypertension from a medical facility.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Change Medication adherence | Patients were assessed Medication adherence at 3 time points: baseline (at the start of the study), 7 months after baseline, and 13 months after baseline
  Medication adherence was assessed using The 8-item Morisky Medication Adherence Scale (MMAS-8). The scale is based on the patients' self-response and consists of eight questions, seven items with yes or no response, and one item with a 5-point Likert scale response option. The total score ranges from 1 to 8, the patient whose adherence score was six or more is considered adherent.

SECONDARY OUTCOMES:
Change Follow-up compliance | Patients were assessed Follow-up compliance at 3 time points: baseline (at the start of the study), 7 months after baseline, and 13 months after baseline
  patients are considered Follow-up compliance when they have had a follow-up examination for hypertension in the past 3 months, according to the doctor's appointment, or early/delayed within 3 days
Change Compliance with reducing salt intake | Patients were assessed Compliance with reducing salt intake at 3 time points: baseline (at the start of the study), 7 months after baseline, and 13 months after baseline
  patients are said to comply with salt reduction when using < 5g salt/day (corresponding to < 1.9g Na/day). Daily sodium intake was calculated based on the Food Frequency Questionnaire (FFQ) on foods high in salt (preserved meat, salt, fish sauce, soy sauce, ketchup) according to the formula [portion size in grams] x [reported consumption frequency (converted to times per day)] x [nutrient per gram]
Change Physical activity compliance | Patients were assessed Physical activity compliance at 3 time points: baseline (at the start of the study), 7 months after baseline, and 13 months after baseline
  Physical activity compliance assessed by The International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF includes 4 questions, collects physical activity information for the previous 7 days regarding vigorous and moderate activity, walking and sedentary behaviors, units in MET-minutes/week. Patients were considered compliant with moderate and high levels of physical activity according to the IPAQ-SF assessment guidelines.
Change Smoking compliance | Patients were assessed Smoking compliance at 3 time points: baseline (at the start of the study), 7 months after baseline, and 13 months after baseline
  patients are considered Smoking compliance when they currently do not smoke or completely quit smoking (including e-cigarettes)
Change Compliance with alcohol consumption | Patients were assessed Compliance with alcohol consumption at 3 time points: baseline (at the start of the study), 7 months after baseline, and 13 months after baseline
  patients are considered Compliance with alcohol consumption when minimizing alcohol consumption, if drinking, the amount should be ≤ 2 standard drinks/day (men) or ≤ 1 standard drinks/day (women), and the total must be ≤ 10 standard drinks/week (men) or ≤ 5 standard drinks/week (women)

CONTACTS AND LOCATIONS:
Locations (1):
- Pham Ngoc Thach University of Medicine, Ho Chi Minh City, Vietnam